CLINICAL TRIAL: NCT05363670
Title: A Phase 2, Single-Dose, Randomized, Active and Placebo Controlled, Four-Period, Cross-Over Study of the Safety and Efficacy of Intranasal Epinephrine After Administration of ARS -1 or Albuterol in Subjects With Persistent Asthma
Brief Title: Administration of ARS-1 or Albuterol in Subjects With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARS Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EPI A01
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 mg/100 µL dose of ARS-1 (Active Comparator)
  Interventions: Drug: ARS-1
- 2 mg/100 µL dose of ARS-1 (Active Comparator)
  Interventions: Drug: ARS-1
- albuterol MDI (180 mcg) (Active Comparator)
  Interventions: Drug: Albuterol MDI
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARS-1 — ARS-1
  Arms: 1 mg/100 µL dose of ARS-1; 2 mg/100 µL dose of ARS-1
Drug: Albuterol MDI — 180 mcg
  Arms: albuterol MDI (180 mcg)
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
ARS-1 is being developed for patients as a needleless alternative route of epinephrine administration for the management of refractory asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 1. Is a male or female subject between the ages of 12 and 65 years, inclusive.
* 2. Asthma that has been stable for at least four weeks prior to screening as defined by clinical history.
* 3. Reversible bronchoconstriction.
* 4. Has body weight more than 30 kilogram (kg) and body mass index between 18 and 34 kg/m², inclusive.
* 5. Has no medical history of hypertension and cardiovascular disease in the last 10 years.
* 6. At screening, has stable vital signs.

Exclusion Criteria:

* 1. History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition.
* 2. Patients receiving beta blocker.
* 3. Has any clinically significant medical condition or physical exam finding as deemed inappropriate by the Investigator.
* 4. Has abnormal cardiovascular exam at screening including any prior history of myocardial infarction or clinically significant abnormal electrocardiogram.
* 5. Has mucosal inflammatory disorders.
* 6. Has had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Effect of ARS-1 versus Albuterol and placebo | From baseline (timepoints 0) to 1 hour
  Difference in forced expiratory volume in 1 second (FEV1) based on area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Tanimoto, MD, PhD, Study Director — ARS Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - University of South Florida, Tampa, Florida
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No